CLINICAL TRIAL: NCT07365709
Title: Liver Cirrhosis Complicated by Clinically Significant Portal Hypertension: the Role of Contrast-enhanced Ultrasound and Splenic Elastography for Non-invasive Assessment
Brief Title: Liver Cirrhosis Complicated by Clinically Significant Portal Hypertension
Acronym: CIRCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pizzolante Fabrizio, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8138
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Portal Hypertension; Spleen Disease; Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Splenic Diseases; Fibrosis | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cirrhosis (Experimental): Adult participants (≥18 years old) with clinically confirmed liver cirrhosis, classified as Child-Pugh class A-C, with clinical and morphological signs of portal hypertension
  Interventions: Drug: SonoVue

INTERVENTIONS:
Drug: SonoVue — microbubbles infusion and ultrasound
  Other Names: INN-sulphur hexafluoride

SUMMARY:
Portal hypertension is a major complication of cirrhosis. HVPG is the diagnostic gold standard but is invasive. Non-invasive tools such as spleen stiffness measurement (SSM) and CEUS show promise for assessing CSPH, though they have not yet been compared directly. A multimodal ultrasound approach may provide a reliable alternative to HVPG.

ELIGIBILITY:
Inclusion Criteria:

Individuals of both sexes aged 18 years or over; Subjects diagnosed with liver cirrhosis. Subjects who have undergone hepatic venous pressure gradient (HVPG) measurement to assess portal hypertension, and/or show indirect clinical signs of significant portal hypertension, such as oesophageal varices or porto-systemic collateral circulation.

Cirrhotic subjects who must undergo contrast-enhanced ultrasound as part of regular hepatological follow-up.

Subjects who have given their informed consent.

Exclusion Criteria:

Subjects aged under 18 years; Subjects with cholestatic disease Subjects diagnosed with clinically significant portal hypertension of non-cirrhotic aetiology.

Subjects diagnosed with ascites Subjects diagnosed with splanchnic thrombosis Subjects presenting with spleno-portal flow reversal Subjects who are allergic to ultrasound contrast media Subjects who have not given their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 12 months
  evaluate the diagnostic performance between the selected parameters and the gold standard for assessing portal hypertension, i.e., HVPG using the ROC curve and calculation of sensitivity, specificity, VPP, VPN, and AUC. Bland-Altman analysis will be applied to assess concordance.

SECONDARY OUTCOMES:
Secondary endpoint | 12 months
  The determination of the ideal cut-off point

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Pizzolante, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: No